CLINICAL TRIAL: NCT07401407
Title: APENERAS: A Prospective Multicenter Observational Study of RICA (ERAS) Pathway Adherence, Safety Outcomes, and Early Discharge Feasibility in Adults Undergoing Urgent Uncomplicated Appendectomy
Brief Title: RICA (ERAS) Pathway Adherence and Early Discharge Feasibility After Urgent Uncomplicated Appendectomy (APENERAS)
Acronym: APENERAS
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Collaborators: Grupo Español de Rehabilitación Multimodal (Other)
Responsible Party: Principal Investigator, Susana Postigo Morales, Staff Anesthesiologist, Hospital Galdakao-Usansolo
Other Study IDs: PI2022120
Record Dates: First submitted 2026-01-14; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Appendicitis; Appendectomy; Ambulatory Surgery
Keywords: ERAS; Enhanced Recovery After Surgery; RICA; urgent surgery; uncomplicated appendicitis; laparoscopic appendectomy; clinical pathway; adherence; early discharge; 30-day outcomes; patient satisfaction; Recuperación intensificada en Cirugía del Adulto
MeSH Terms: conditions — Appendicitis; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urgent Uncomplicated Appendectomy Cohort: Adults undergoing urgent laparoscopic appendectomy for uncomplicated acute appendicitis in participating hospitals. Perioperative management follows routine clinical practice. The adherence to the RICA (ERAS) pathway items is assessed, along with safety outcomes and early discharge feasibility.

SUMMARY:
This multicenter, prospective observational study (APENERAS) evaluates adherence to the RICA (ERAS Zaragoza 2022) perioperative care pathway in adults undergoing urgent laparoscopic appendectomy for uncomplicated acute appendicitis. The study aims to describe real-world adherence to the pathway across participating hospitals and to explore its association with patient safety and recovery outcomes.

Key outcomes include postoperative complications (including severity), length of hospital stay, and readmissions within 30 days. Patient-reported satisfaction is also assessed using a structured survey. In addition, the study evaluates the feasibility of early discharge/ambulatory management by intention-to-treat, using a standardized checklist of clinical, functional, and social discharge criteria assessed during the first 24 hours after surgery.

No changes to usual clinical care are introduced. Data are collected from routine perioperative management and follow-up.

DETAILED DESCRIPTION:
APENERAS is a prospective, multicenter observational study conducted in adult patients undergoing urgent laparoscopic appendectomy for uncomplicated acute appendicitis. The study assesses real-world adherence to the RICA (ERAS Zaragoza 2022) pathway, a structured set of perioperative recommendations intended to optimize recovery and standardize care in urgent surgery settings.

The primary objective is to quantify overall adherence and adherence by individual components of the pathway. Secondary objectives include evaluating the association between adherence and (1) postoperative safety outcomes (complications and severity classification), (2) efficiency outcomes (length of stay), (3) unplanned healthcare use (readmissions within 30 days), and (4) patient experience (satisfaction survey completed at discharge). In addition, feasibility of early discharge/ambulatory management is assessed by intention-to-treat using a standardized discharge-readiness checklist (clinical stability, pain control with oral analgesia, oral tolerance, mobilization, spontaneous urination, wound status, and social support), evaluated during the first postoperative day.

Candidate profiles for early discharge are also explored using established clinical prediction tools (e.g., Saint-Antoine Score), together with demographic and clinical covariates. Follow-up is performed up to 30 days after surgery to capture postoperative events and readmissions.

This study does not involve any experimental intervention, drug, or device, and does not require changes to standard clinical practice. It is based on systematic data collection from routine care processes and clinical records in each participating center.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years.
* Immunocompetent patients.
* ASA physical status I-III.
* Preoperative diagnosis of uncomplicated acute appendicitis (based on clinical assessment, laboratory tests, and imaging such as ultrasound and/or CT according to availability).
* Indication for urgent appendectomy for uncomplicated appendicitis.
* Laparoscopic approach.
* Expected operative time < 90 minutes.
* Cooperative patient able to understand and follow instructions.
* Voluntary participation and written informed consent.
* Adequate social/family support (availability of a responsible adult for transport home and support during the first postoperative days).
* Travel time from home to hospital < 1 hour and access to transportation.
* Acceptable home environment for recovery (telephone access and basic habitability/hygiene).

Exclusion Criteria:

* ASA physical status IV.
* Age < 18 years or > 75 years.
* BMI > 35 kg/m² with significant respiratory or cardiovascular complications.
* Ischemic heart disease class IV or acute myocardial infarction within the last 6 months.
* Congestive heart failure NYHA class III-IV.
* Sleep apnea or severe COPD, or need for home oxygen therapy.
* Poorly controlled diabetes mellitus.
* Severe psychiatric disorders, drug addiction, or severe alcoholism.
* History of major anesthesia-related complications or malignant hyperthermia.
* Epilepsy.
* Pregnancy.
* Use of anticoagulants, MAO inhibitors, systemic corticosteroids, or immunosuppressive drugs.
* Complicated appendicitis (gangrenous or perforated appendicitis, abscess, diffuse peritonitis).
* Severe sepsis.
* Primary open appendectomy or conversion to open surgery.
* Positive SARS-CoV-2 PCR or symptoms compatible with COVID-19.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-75 years undergoing urgent laparoscopic appendectomy for uncomplicated acute appendicitis in participating hospitals. The study evaluates adherence to the RICA (ERAS Zaragoza 2022) pathway in routine clinical practice, early discharge feasibility (8, 12, and 24 hours after surgery), and safety outcomes (complications, readmissions, reinterventions, and mortality) up to 30 days after surgery. No experimental intervention is introduced.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Overall adherence to the RICA (ERAS Zaragoza 2022) pathway | From day of surgery through postoperative day 2 or hospital discharge (whichever occurs first).
  Overall adherence will be quantified as the proportion (%) of prespecified RICA (ERAS Zaragoza 2022) items fulfilled per participant and overall, using the study case report form. Adherence will be reported as a global percentage and by individual pathway components.

SECONDARY OUTCOMES:
Early discharge feasibility at 8, 12 and 24 hours after surgery | 8, 12 and 24 hours after surgery.
  Feasibility of early discharge will be assessed by intention-to-treat using a standardized discharge-readiness checklist (clinical stability, respiratory stability, orientation, mobility, oral intake, urination, wound status, and social support/logistics). The proportion of patients meeting all criteria at each timepoint (8h, 12h, 24h) will be reported.
Postoperative complications and severity (Clavien-Dindo) | Up to 30 days after surgery.
  Postoperative complications will be recorded and graded according to the Clavien-Dindo classification.
Length of hospital stay | Time from surgery (Day 0) to hospital discharge (index hospitalization); assessed at discharge (followed until discharge, up to 30 days post-surgery).
  Length of stay will be measured as time from surgery to hospital discharge (reported in days and/or hours as available).
Readmission within 30 days | Up to 30 days after discharge.
  Unplanned readmissions for any cause will be recorded.
Patient satisfaction score | Up to 30 days after surgery.
  Patient satisfaction will be assessed using a structured survey delivered at hospital discharge and collected during postoperative follow-up. The overall satisfaction score (0-10 scale) and relevant domains will be analyzed.
Saint-Antoine Score for early discharge eligibility prediction within 24 hours after surgery | Baseline (preoperative; assessed immediately before surgery).
  The Saint-Antoine Score is a 5-point preoperative clinical score (range: 0 to 5) calculated at baseline (immediately before surgery) as the sum of five low-risk criteria (each criterion = 1 point; total score 0-5). Higher scores indicate a greater likelihood of eligibility for unplanned early discharge within 24 hours (better discharge readiness/lower-risk profile). Lower scores indicate a lower likelihood of early discharge eligibility. Predictive performance will be described (e.g., proportion eligible across score categories and discrimination metrics, as applicable).
Reintervention within 30 days | Up to 30 days after surgery.
  Any unplanned reintervention after the index appendectomy, including surgical reoperation (e.g., re-laparoscopy/laparotomy) and other invasive procedures (e.g., percutaneous drainage), will be recorded.
All-cause mortality within 30 days | Up to 30 days after surgery.
  All-cause mortality will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bakarne Ugarte-Sierra, PhD, Study Director — Grupo español de rehabilitación multimodal (GERM); José Manuel Ramírez-Rodríguez, PhD, Study Director — Grupo español de rehabilitación multimodal (GERM)
Locations (4):
- Spain (4):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari d'Igualada, Igualada, Barcelona
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in publications will be shared. The shared dataset will contain coded study IDs and will exclude direct identifiers (e.g., name, medical record number, address). Variables will be minimized/modified as needed to reduce re-identification risk in accordance with GDPR and institutional policies.
Supporting Information: Study Protocol, SAP
Time Frame: Available beginning 12 months after publication of the primary results and for 5 years thereafter.
Access Criteria: Access will be granted to researchers with a clear research question and an appropriate analysis plan, subject to review and approval by the study team and compliance with GDPR and applicable institutional policies. Data will be provided in de-identified form after completion of a data sharing agreement. Requests should be submitted by email to: estudioapeneras@gmail.com

REFERENCES:
- [Background] Postigo-Morales S, Ugarte-Sierra B, San-Juan-Gonzalez M, Ramirez-Rodriguez JM. [Implementation of the ERAS pathway in emergency surgery: adherence, barriers and facilitators]. J Healthc Qual Res. 2025 Oct 31;41(1):101170. doi: 10.1016/j.jhqr.2025.101170. Online ahead of print. Spanish. PMID 41175821
- [Background] Scott MJ, Aggarwal G, Aitken RJ, Anderson ID, Balfour A, Foss NB, Cooper Z, Dhesi JK, French WB, Grant MC, Hammarqvist F, Hare SP, Havens JM, Holena DN, Hubner M, Johnston C, Kim JS, Lees NP, Ljungqvist O, Lobo DN, Mohseni S, Ordonez CA, Quiney N, Sharoky C, Urman RD, Wick E, Wu CL, Young-Fadok T, Peden CJ. Consensus Guidelines for Perioperative Care for Emergency Laparotomy Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations Part 2-Emergency Laparotomy: Intra- and Postoperative Care. World J Surg. 2023 Aug;47(8):1850-1880. doi: 10.1007/s00268-023-07020-6. Epub 2023 Jun 5. PMID 37277507
- [Background] Raimbert P, Voron T, Laroche S, O'Connell L, Debove C, Challine A, Parc Y, Lefevre JH. Ambulatory appendectomy for acute appendicitis: Can we treat all the patients? A prospective study of 451 consecutive ambulatory appendectomies out of nearly 2,000 procedures. Surgery. 2023 May;173(5):1129-1136. doi: 10.1016/j.surg.2023.01.003. Epub 2023 Feb 10. PMID 36775758
- [Background] Gignoux B, Blanchet MC, Lanz T, Vulliez A, Saffarini M, Bothorel H, Robert M, Frering V. Should ambulatory appendectomy become the standard treatment for acute appendicitis? World J Emerg Surg. 2018 Jun 28;13:28. doi: 10.1186/s13017-018-0191-4. eCollection 2018. PMID 29988464
- [Background] Ruiz-Tovar J, Llavero C, Perez-Lopez M, Garcia-Marin A. Implementation of an Enhanced Recovery After Surgery (ERAS) protocol for acute complicated and uncomplicated appendicitis. Tech Coloproctol. 2021 Sep;25(9):1073-1078. doi: 10.1007/s10151-021-02484-x. Epub 2021 Jun 26. PMID 34173925
- [Background] Trejo-Avila ME, Romero-Loera S, Cardenas-Lailson E, Blas-Franco M, Delano-Alonso R, Valenzuela-Salazar C, Moreno-Portillo M. Enhanced recovery after surgery protocol allows ambulatory laparoscopic appendectomy in uncomplicated acute appendicitis: a prospective, randomized trial. Surg Endosc. 2019 Feb;33(2):429-436. doi: 10.1007/s00464-018-6315-9. Epub 2018 Jul 9. PMID 29987566
- [Background] Di Saverio S, Podda M, De Simone B, Ceresoli M, Augustin G, Gori A, Boermeester M, Sartelli M, Coccolini F, Tarasconi A, De' Angelis N, Weber DG, Tolonen M, Birindelli A, Biffl W, Moore EE, Kelly M, Soreide K, Kashuk J, Ten Broek R, Gomes CA, Sugrue M, Davies RJ, Damaskos D, Leppaniemi A, Kirkpatrick A, Peitzman AB, Fraga GP, Maier RV, Coimbra R, Chiarugi M, Sganga G, Pisanu A, De' Angelis GL, Tan E, Van Goor H, Pata F, Di Carlo I, Chiara O, Litvin A, Campanile FC, Sakakushev B, Tomadze G, Demetrashvili Z, Latifi R, Abu-Zidan F, Romeo O, Segovia-Lohse H, Baiocchi G, Costa D, Rizoli S, Balogh ZJ, Bendinelli C, Scalea T, Ivatury R, Velmahos G, Andersson R, Kluger Y, Ansaloni L, Catena F. Diagnosis and treatment of acute appendicitis: 2020 update of the WSES Jerusalem guidelines. World J Emerg Surg. 2020 Apr 15;15(1):27. doi: 10.1186/s13017-020-00306-3. PMID 32295644
- See also: GERM - Protocolos Zaragoza (RICA/ERAS) - Urgencias: Uncomplicated Acute Appendicitis — https://grupogerm.es/protocolos-zaragoza/